CLINICAL TRIAL: NCT04896671
Title: Neural Mechanism of Physical Exercise in Enhancing Executive and Social Functions in Adolescents
Brief Title: Physical Exercise Training to Enhance Executive and Social Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other); Griffith University (Other)
Responsible Party: Principal Investigator, LAM, Yin Hung, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20190311003
Record Dates: First submitted 2020-10-15; First posted 2021-05-21 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Broad Autism Phenotype
Keywords: physical exercise; social function; broad autism phenotype; executive function
MeSH Terms: conditions — Motor Activity; Social Adjustment | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A total of 30 participants with BAP were randomly assigned to either groups: 1) intervention group (12 treadmill running sessions, two sessions per week and each session 30 minutes) and 2) control group: waitlist control group.
Who Masked: Participant
Masking Description: The participants would not know there are two groups. Each participant would assume to participate in physical exercise at some point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Each participant joins a total of 12 treadmill running sessions, two sessions per week and each session for 30 minutes.
  Interventions: Behavioral: Physical exercise (running on a treadmill)
- Waitlist control group (No Intervention): They receive no treatments.

INTERVENTIONS:
Behavioral: Physical exercise (running on a treadmill) — Participants in the intervention group join a total of 12 treadmill running sessions, two sessions per week and each session for 30 minutes. In each session, every participant will be trained to run for 30 minutes on a treadmill. According to Exercise and Sports Science Australia (ESSA) exercise intensity guidelines, the intensity of running is suggested to be moderate and vigorous (alternating between the two) in this study.
  Arms: Intervention group

SUMMARY:
Background and study aims: Executive functions (EF) and social functions are important for self-regulation, problem solving, and attaining future goals yet they are impaired in Autism Spectrum Disorder (ASD). Physical exercise (PE) is found to enhance these central cognitive and social impairments in ASD. While limited research has begun to target these impairments in clinical samples, the presence of sub-clinical traits of ASD (refer to as broad autism phenotype (BAP)) in the general population is more common than the 1% prevalence of ASD. Therefore, it is crucial to study these impairments in the sub-clinical individuals. This study aims to investigate the effectiveness of PE in enhancing the EF and social functions in the BAP adolescents. Method: Participants will be recruited from the local community and they should be between the age of 7-20 years without any psychiatric disorders. Expected results: PE is predicted to be effective in reducing the EF and social impairments in these adolescents. Implications: These findings can inform us with the knowledge to design a community-based PE training targeting EF problems in these adolescents with BAP in the local context. Ultimately, this training can be incorporated to the curriculum of the primary and secondary schools targeting BAP and associated impairments in adolescents.

DETAILED DESCRIPTION:
Executive functions (EF) refer to goal-directed cognitive processes consisting of three major components including cognitive flexibility (mental flexibility), inhibition (inhibitory control) and working memory. These components interact with each other and play a crucial role in a range of life outcomes including mental and physical health, school and job success and marital harmony. In addition, higher EF is associated with better problem solving, reasoning and planning skills as well as social functions.

Autism spectrum disorder (ASD) is a neurodevelopmental disorder characterised by social communication and interaction impairments, as well as restricted and repetitive patterns of behavior. Individuals with ASD have EF impairments which are linked to the restricted and repetitive behaviors that characterise this condition. The prevalence of ASD is increasing with as many as 1 in 68 individuals, which further augments the burden to the ASD individuals, their families and society. Hence, it is essential to investigate the underlying mechanism of ASD and design a cost-effective training that can be widely adopted in the community to reduce impairments arising from ASD symptoms.

Importantly, ASD traits occur on a continuum, and increasingly there is recognition of a broader autism phenotype (BAP) in those that show sub-clinical symptoms. Similarly, these individuals also show impairments in executive function and social functions, making this group an important target for the development and implementation of interventions. As such, we can deliver appropriate training at an earlier stage to prevent associated impairments in those with ASD traits. Therefore, instead of ASD, the present study examines the individuals with BAP.

Given EF impairments along with social function deficits are found in the sub-clinical individuals with BAP, is the training pertaining to ASD applicable to these individuals? In prior literature, physical exercise (PE) has been proved to enhance EF and social functions. For instance, regular PE can enhance cerebral blood flow and increase the formation of new blood vessels in a number of brain regions that are involved in EF and social functions. More specifically, PE is shown to enhance the performance of EF in healthy children and pre-adolescents and those with ASD. For example, it was found that PE including jogging significantly decreased the repetitive and off-task behaviors and the level of aggression in individuals with ASD. Nevertheless, although PE is shown to be beneficial to reduce the symptoms and EF as well as social impairments in ASD, whether it produces the same positive outcomes in the non-clinical individuals. To address the research questions listed above, this proposed study aims to investigate whether PE training enhances the EF and social functions in the adolescents with BAP.

Although the benefits of physical exercise have been studied in the ASD, BAP is under studied in prior literature. This proposed study will extend from the current literature to investigate the non-clinical group who have autistic traits with a longitudinal and randomized controlled trial design (RCT). The findings of this proposed study have multiple levels of significance and implications. For instance, if the hypotheses are supported, the PE training which is more cost-effective than psychotherapy in treating EF and social functioning deficits and associated impairments can be promoted to school settings. Ultimately, it can be incorporated to the curriculum of the primary and secondary schools to reduce BAP and associated impairments in the adolescents. Secondly, by examining those with sub- clinical symptoms, this research will contribute to early trainings approaches for the condition. Lastly, this proposed study can also help promote physical activities among adolescents which can further decrease mental and health issues in the local context.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 7 to 20
* Studying at one of the local schools
* Have never been diagnosed with ASD or any other disorder listed in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* Are not currently under any psychiatric medications or therapies

Exclusion Criteria:

* Have been diagnosed with ASD or any other disorder listed in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* Are currently under any psychiatric medications or therapies

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Based on born gender.
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Demographics | Before intervention (baseline)
  A simple demographic questionnaire will be used to gather participants personal information, including age, gender, current medication or therapy, and medical history of the participant and his/her family members.
Change from baseline autistic traits at 6 weeks | baseline and 6- week follow up
  The Autism-Spectrum Quotient-Adolescent Version (AQ-Adolescent; Baron-Cohen et al., 2006) and related self-report scales will be used to measure ASD traits. The AQ- adolescent is a self-report questionnaire comprising of 50 items assessing five areas, namely social, attention switching, attention to detail, communication and imagination.
Change from baseline executive functions at 6 weeks | baseline and 6- week follow up
  EF and social functions will be measured using the Cambridge Neuropsychological Test Automated Battery (CANTAB). The CANTAB is a computerized test battery targeting multiple neuropsychological functions. This battery includes Reaction Time, Paired Associates Learning, Spatial Working Memory, One Touch Stockings of Cambridge, Multitasking Test, and Emotion Recognition Task.
Change from baseline psychological resilience at 6 weeks | baseline and 6- week follow up
  Participant's psychological resilience will be measured by 10-item Connor-Davidson Resilience Scale (CD-RISC).
Change from baseline schizotypal personality traits at 6 weeks | baseline and 6- week follow up
  Schizotypal Personality Questionnaire will be used to measure schizotypal personality traits.

SECONDARY OUTCOMES:
Change from baseline aggression at 6 weeks | baseline and 6- week follow up
  Reactive and Proactive Aggression Questionnaire will be used to measure aggression in the participants.
Change from baseline empathy at 6 weeks | baseline and 6- week follow up
  Cognitive, Affective and Somatic Empathy Scale (CASES) will be used to measure empathy.

CONTACTS AND LOCATIONS:
Overall Officials: Bess Yin-Hung Lam, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

DOCUMENTS (3):
  • Study Protocol (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT04896671/Prot_003.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT04896671/SAP_004.pdf
  • Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT04896671/ICF_005.pdf